CLINICAL TRIAL: NCT07113210
Title: Understanding Quality of Life in Presbyopic Patients Who Are Treated With Qlosi
Brief Title: Quality of Life in Presbyopic Patients Who Are Treated With Qlosi
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Southern College of Optometry (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: qlosi00006733
Record Dates: First submitted 2025-08-02; First posted 2025-08-08 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Presbyopia; Glasses; Dry Eye
MeSH Terms: conditions — Presbyopia; Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Participant's who qualify will be given Qlosi and instructions for how many drops to take.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Qlosi (Experimental): Subjects will be treated with Qlosi™ BID OD/OS, and subjects will only be allowed to use reading glasses for urgent work
  Interventions: Drug: pilocarpine HCL ophthalmic solution

INTERVENTIONS:
Drug: pilocarpine HCL ophthalmic solution — Qlosi will be given to participants and quality of life will be determined.

SUMMARY:
The goal of this clinical trial is to determine how Qlosi™ (pilocarpine HCL ophthalmic solution) 0.4%impacts the quality of life of participants with presbyopia by using a battery of validated and investigator-developed instruments

* Improvement in presbyopic symptoms as measured with the Near Activity Visual Questionnaire-Presbyopia (NAVQ-P) when using Qlosi™ at week 4 compared to baseline (continuous variable).
* Improvement in presbyopic symptoms as measured with the Visual Quality of Life with Time Survey (VisQualT) questionnaire when using Qlosi™ at week 4 compared to baseline.

DETAILED DESCRIPTION:
This will be a prospective, multi-center, study. Subjects will be treated with Qlosi™ BID OD/OS, and subjects will only be allowed to use reading glasses for urgent work. All subjects will be prescribed a pair of distance spectacles (no near add) at the screening visit. The baseline survey and visual acuity data will be collected at the spectacle dispense visit (outcome measures). The screening visit data will be used as the baseline data for slit-lamp biomicroscope and indirect ophthalmoscopy and not repeated at the dispense visit. The investigators feel that this approach is reasonable because it is unlikely that the slit-lamp biomicroscope and indirect ophthalmoscopy data will change between the screening visit and dispense visit. Distance spectacles will be provided at a dispense visit 1-2 weeks after screening and a logMAR visual acuity of 0.00 or better OD/OS at distance will be confirmed. Subjects will then be instructed to start their treatment. After 4 weeks, subjects will return for an evaluation visit that will occur 4-6 hours after starting treatment for the day. Subjects will then be compensated for their time and exited from the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are 45-64 years old (inclusive) at the time of screening.
* Be able and willing to provide written informed consent and sign a Health Information Portability and Accountability Act (HIPAA) form prior to any study procedure being performed.
* Be able and willing to follow all instructions and attend study visits.
* Have text messaging capabilities on their phone.
* Self-reported complaints of near vision blur when fully corrected at distance.
* Study confirmed near add that is between +0.75 D to +2.00 D OD/OS (inclusive).
* Spherical distance prescription between +1.00 D to -4.00 D OD/OS (inclusive).
* Cylinder power less than or equal to -1.00 D OD/OS.
* Best-corrected visual acuity (BCVA) at distance of 0.00 logMAR (20/20 Snellen equivalent) or better OD/OS.

Exclusion Criteria:

* Known hypersensitivity to any ingredient in the study drops.
* Any active ocular condition that may confound study results (e.g., dry eye, allergy, conjunctivitis, ocular infection).
* Any use of prescription eye drops 1 week before screening or during the study.
* Any past use of the study drops.
* Any contact lens use for the duration of the study.
* Artificial tears or lubricant eye drops use on the day of or during any study visits.
* Clinically significant abnormal findings (e.g., central corneal scar) on a slit lamp exam in either eye documented at screening or a known history of a clinically significant slit-lamp finding in either eye that could confound study results.
* Have had an ocular surgical intervention within 6 months of the screening visit or planned surgical intervention during the study.
* A female of childbearing potential who is currently pregnant, nursing, or planning a pregnancy.
* Any visible retinal findings noted upon a dilated fundus examination known to be a risk for use of study treatment (as determined by the investigator).

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Near Visual Acuity Questionnaire-Presbyopia | 1 month
  • Improvement in presbyopic symptoms as measured with the Near Activity Visual Questionnaire-Presbyopia (NAVQ-P) when using Qlosi at week 4 compared to baseline (continuous variable). In which higher scores are better.

SECONDARY OUTCOMES:
Visual Quality of Life with Time Survey (VisQualT) | 1 month
  • Improvement in presbyopic symptoms as measured with the Visual Quality of Life with Time Survey (VisQualT) questionnaire when using Qlosi™ at week 4 compared to baseline
Improvement in overall visual acuity score | 1 month
  • Improvement in presbyopic symptoms as measured with the overall quality of life VAS when using Qlosi™ at week 4 compared to baseline. In which higher scores are better
Investigator developed survey | 1 month
  • Improvement in presbyopic symptoms as measured with the Investigator-Developed Likert Survey when using Qlosi at week 4 compared to baseline. In which positive answers such as strongly agree are better.
Text message surveys | 1 day, 1 week, 1 month
  • Real-time text messaging to subjects on each day of treatment to identify time to treatment onset post-drop application (minutes). In which lower scores are better.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Complete Eye Care of Medina, Medina, Minnesota
  - The Southern College of Optometry, Memphis, Tennessee